CLINICAL TRIAL: NCT01934920
Title: Identifying Patients With Unrecognized Treatable Diabetic Macular Edema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Elman Retina Group (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Elman-01
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This trial will assess the incidence of new and/or undiagnosed diabetic macular edema (DME) in diabetic patients that undergo a DME screening exam. The screening exam will consist of medical history, Electronic ETDRS visual acuity assessment, SD-OCT and color fundus photography

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Patient related considerations
* Patients with diabetes mellitus
* Disease related considerations
* Diabetes mellitus

Exclusion Criteria:

* Prior admission screening within twelve months.
* Inability to sit for evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients identified through medical records or admitted into Franklin Square Hospital with a history of diabetes
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Assess the incidence of new and/or undiagnosed diabetic macular edema. | 1 day (Patients are only seen once for assessments)
  This trial will assess the incidence of new and/or undiagnosed diabetic macular edema (DME) in diabetic patients that undergo a DME screening exam. The screening exam will consist of medical history, Electronic ETDRS visual acuity assessment, SD-OCT and color fundus photography

SECONDARY OUTCOMES:
Streamlining and identification of patients at risk of diabetic macular edema | 1 day (Patients only seen once for assessments)
  Establish methods for streamlining screening and identification of patients at risk.
  Establish methods for referral for treatment of patients identified with vision threatening diabetic retinopathy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Elman, MD, Principal Investigator — Elman Retina Group, P.A.
Locations (2):
- United States (2):
  - Aaron Goldberg, Primary Care, Baltimore, Maryland
  - MedStar Hospital, Baltimore, Maryland